CLINICAL TRIAL: NCT02789046
Title: DIFFICULT PERIPHERAL INTRAVENOUS ACCESS IN ADULT DURING THE PREOPERATIVE PERIOD
Brief Title: DIFFICULT INTRAVENOUS ACCESS IN ADULTS (VENSCORE)
Acronym: VENSCORE
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBXSAR32016-01
Record Dates: First submitted 2016-05-24; First posted 2016-06-02 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-03

CONDITIONS: Peripheral Venous Catheterization
Keywords: adult; vascular access; preoperative period; peripheral venous catheterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: peripheral intravenous catheterization — success or failure intravenous placement on first attempt and factors associated with failed intravenous catheterization

SUMMARY:
The objective of the prospective multicenter observational study consists in defining a difficult intravenous access score in adult, during the preoperative period.

The main objective: the outcome of interest is defined as failure of cannulation on first attempt.

The risk factors of failure of cannulation on first attempt will be described. Adjusted multivariate models will be constructed. A prediction model will be proposed according to the transparent reporting of a multivariable prediction model for individual prognosis or diagnosis (TRIPOD)

DETAILED DESCRIPTION:
Objectives:

To define a difficult intravenous access score in adult during the preoperative period Methods Multicenter, Observational prospective study

Patients:

patients >18 years old, undergoing peripheral IV placement just before a surgery in operating room excision criteria: pregnant woman, induction of anesthesia with sevoflurane, Predictor variables include: history of patient (age,BMI, Fitzpatrick skin type, cancer, ICU stay, burn, diabetes, kidney disease, anxiety of patient...) , operator experience characteristics( years since graduation, years of anesthesiology experience, IVs started per month), type of catheter and place of catheterization),and postcatheterization data (success on fist attempt yes or no, number of total attempts until success...)

ELIGIBILITY:
Inclusion Criteria:

* patients >18 years old, undergoing peripheral IV placement just before a surgery in operating room

Exclusion Criteria:

* patients who refused IV placement; pregnant woman; induction of anesthesia with sevoflurane without venous access in place

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing peripheral intravenous placement just before a surgery will be enrolled. (the investigator does not assign specific interventions to the subjects of the study)
Sampling Method: Non-Probability Sample
Enrollment: 3300 (Actual)
Dates: Start 2016-06; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
failure intravenous placement on the first attempt | during the hour before surgery

SECONDARY OUTCOMES:
risk factors associated with failure intravenous catheterization | during the hour before surgery

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - Centre Hospitalier Sud Gironde, Lagon, France
  - CHU Saint Pierre, Saint Pierre La Réunion, Ile de La Réunion
  - Centre Hospitalier d'Agen, Agen
  - Centre Médico-chirurgical Wallerstein, Arès
  - Centre Hospitalier de la Cote Basque, Bayonne
  - Clinique Saint Augustin Bordeaux, Bordeaux
  - Institut Bergonié, Bordeaux
  - Centre hospitalier Universitaire de Bordeaux, Bordeaux
  - Hôpital d'instruction des Armées Robert Picqué, Bordeaux
  - Centre Hospitalier de Dax, Dax
  - Centre Hospitalier d'Arcachon, La Teste-de-Buch
  - Centre Hospitalier de Libourne, Libourne
  - Centre Hospitalier de Mont de Marsan, Mont-de-Marsan
  - Centre Hospitalier de Pau, Pau
  - Centre Hospitalier de Périgueux, Périgueux
  - Centre Hospitalier de Tahiti, Tahiti